CLINICAL TRIAL: NCT01909973
Title: Mobile Technology to Engage and Link Patients and Providers in Antidepressant Treatment
Acronym: Medlink RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Director, Center for Behavioral Intervention Technologies; Professor, Department of Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH095907-02-RCTML; R34MH095907-02 (NIH); NCT01583764 (obsolete NCT alias)
Record Dates: First submitted 2013-07-17; First posted 2013-07-29 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Depression
Keywords: Depression; Antidepressant Medication; Adherence; Mobile Smartphone Intervention; Telemedicine; Primary Care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MedLink System (Experimental): For 12 weeks, the patient who is newly prescribed antidepressant medication will receive a mobile phone and a GSM enable pill bottle in order to provide and receive feedback regarding medication adherence.
  Interventions: Behavioral: MedLink System
- Treatment As Usual (No Intervention): Patients will continue to receive treatment as usual from their primary care doctor. Patients in this arm will also receive a free mobile phone for the 12 weeks of the intervention.

INTERVENTIONS:
Behavioral: MedLink System — Patient adherence to anti depressant medication will be accomplished by 1) monitoring adherence and providing feedback to patient (e.g. prompting patient to take medication); 2) monitoring side effects and treatment response and providing in-the-moment feedback and support; 3) activating the patient to take appropriate action (e.g. call the prescribing physician) based upon monitoring data; 4) providing standardized education and positive reinforcement to the patient.
  The care team will be supported and activated by being provided 1) suggested guideline-congruent actions and 2) timely information regarding the patient's status.
  Arms: MedLink System

SUMMARY:
The goal of this project is to develop and pilot a mobile smartphone delivered intervention that will improve antidepressant medication care by providing medication adherence monitoring and support to the patient, feedback on patient adherence and response to treatment to the primary care team, and information to both patients and providers on guideline-congruent care personalized to the patient's response to antidepressant medication.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is common and imposes a very high societal burden in terms of cost, morbidity, suffering, and mortality. While primary care is the de facto site for treatment of MDD, outcomes in primary care are poor. Two principal reasons for the poor outcomes in primary care are poor patient adherence to antidepressant medications (ADMs) and the failure of physicians to provide guideline-congruent care. This problem is aggravated by a lack of communication between patients and the care team.

A growing body of research indicates that primary care-centered strategies aimed at enhancing guideline-congruent care have not been effective. Interventions aimed at improving adherence in the patient have been successful in changing patient adherence behavior; however these frequently fail to improve depression outcomes, particularly when there is no intervention on the physician side to encourage optimization of ADMs. Recent developments in information and communications technologies (ICT) have opened new opportunities to improve health and mental health care, and to link patients and their providers. This study harnesses these advances to develop and pilot a system where ADM adherence will be passively measured using an electronic pill dispenser. The dispenser is connected to a mobile smartphone via Global System for Mobile Communications (GSM), so that targeted, timely reminders can be provided when the patient fails to take the ADM. When the patient is adherent, the patient will not be bothered with reminders. Depressive symptoms and side-effects will be periodically monitored weekly via the phone. Every 4 weeks, or if indicated (e.g intolerable side effects or urgent situations), primary care teams will receive notifications via the electronic medical record that include a summary of patient data on treatment response and side effects, guideline-congruent treatment recommendations based on patient data and a recommendation to contact the patient, if indicated. Simultaneously, a similar message will be provided to the patient via short message service (or text), including feedback, possible treatment options, and a recommendation to contact the physician's office. Thus, both the patient and care team will be activated to provide, request and adhere to guideline-congruent care.

The aim of this study is to develop and pilot the medLink system. Development will employ an iterative user-centered approach. The pilot trial will compare 12 weeks of the medLink system to a treatment as usual control among primary care patients with MDD initiating ADM treatment. Outcomes will include patient adherence to ADM, physician adherence to treatment guidelines, and depression.

ELIGIBILITY:
Inclusion Criteria:

* Has been prescribed an antidepressant medication by a Primary Care Provider, but has not yet initiated treatment
* Has depression determined by primary care physician
* Is familiar with the use of mobile phones
* Is able and willing to carry the mobile phone
* Is able to speak and read English
* Is at least 18 years of age

Exclusion Criteria:

* Is current taking an antidepressant medication or has taken one in the previous 3 months
* Has visual, hearing, voice, or motor impairment that would prevent completion of study procedures or use of mobile phone
* Is diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, current substance dependence, or other diagnosis for which participation in this trial is either inappropriate or dangerous. Patients with substance dependence diagnoses who have been clean and sober for 12 months will be admitted if otherwise eligible
* Is severely suicidal (has ideation, plan, and intent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Northwestern Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MedLink System: For 12 weeks, the patient who is newly prescribed antidepressant medication will receive a mobile phone and a GSM enable pill bottle in order to provide and receive feedback regarding medication adherence.
  MedLink System: Patient adherence to anti depressant medication will be accomplished by 1) monitoring adherence and providing feedback to patient (e.g. prompting patient to take medication); 2) monitoring side effects and treatment response and providing in-the-moment feedback and support; 3) activating the patient to take appropriate action (e.g. call the prescribing physician) based upon monitoring data; 4) providing standardized education and positive reinforcement to the patient.
  The care team will be supported and activated by being provided 1) suggested guideline-congruent actions and 2) timely information regarding the patient's status.
Period: Overall Study
Arm/Group | MedLink System | Treatment As Usual
Started | 8 | 7
Completed | 7 | 7
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MedLink System | Treatment As Usual | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (17.04) | 42.3 (14.02) | 46 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Antidepressant Medication
Description: Frequency of medication usage from baseline to end of treatment
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | MedLink System | Treatment As Usual
Number analyzed (Participants) | 8 | 7
Participants
  Baseline: 01. Missed med in last 2 wks? - missed all 14 days | 0 | 0
  Baseline: 01. Missed med in last 2 wks? - missed 6 to 8 days | 0 | 1
  Baseline: 01. Missed med in last 2 wks? - missed 3 to 5 days | 0 | 1
  Baseline: 01. Missed med in last 2 wks? - missed once/twice | 2 | 1
  Baseline: 01. Missed med in last 2 wks? - No, took every day | 6 | 4
  Baseline: 02a. Stopped med during last 2 wks? - Yes | 0 | 0
  Baseline: 02a. Stopped med during last 2 wks? - No | 8 | 7
  Baseline: 2aii. Stopped meds due to: Side effects - Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 2aii. Stopped meds due to: Symptoms increase -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 2aii. Stopped meds due to: Symptoms decrease -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 2aii. Stopped meds due to: Ran out of meds -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 2aii. Stopped meds due to: Forgot to take -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02b. Skipped med in last 2 wks? - Yes | 1 | 0
  Baseline: 02b. Skipped med in last 2 wks? - No | 7 | 7
  Baseline: 02bi. Skipped meds due to: Side effects - Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02bi. Skipped meds due to: Symptoms increase -Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02bi. Skipped meds due to: Symptoms decrease -Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02bi. Skipped meds due to: Ran out of meds -Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02bi. Skipped meds due to: Forgot to take -Yes | 1 | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02bi. Skipped meds due to: Other reason -Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02c. Have you reduced med dosage? - Yes | 0 | 0
  Baseline: 02c. Have you reduced med dosage? - No | 8 | 7
  Baseline: 02ci. Reduced meds due to: Side effects - Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02ci. Reduced meds due to: Symptoms increase -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02ci. Reduced meds due to: Symptoms decrease -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02ci. Reduced meds due to: Ran out of meds -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02ci. Reduced meds due to: Forgot to take -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02ci. Reduced meds due to: Other reason -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02d. Have you increased med dosage? - Yes | 1 | 1
  Baseline: 02d. Have you increased med dosage? - No | 7 | 6
  Baseline: 02di. Increased meds due to: Side effects - Yes | 0 | 0
  Baseline: 02di.Increased meds due to: Symptoms increase -Yes | 0 | 0
  Baseline: 02di.Increased meds due to: Symptoms decrease -Yes | 0 | 0
  Baseline: 02di.Increased meds due to: Ran out of meds -Yes | 0 | 0
  Baseline: 02di.Increased meds due to: Forgot to take -Yes | 0 | 0
  Baseline: 02di.Increased meds due to: Other reason -Yes | 1 | 1
  Baseline: 02ai. Stopped meds 3 days ago | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02ai. Stopped meds 14 days ago | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Baseline: 02ai. Stopped meds 2 ± 0 days days ago | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 4: 01. Missed med in last 2 wks? - missed all 14 days | 0 | 0
  Week 4: 01. Missed med in last 2 wks? - missed 6 to 8 days | 0 | 1
  Week 4: 01. Missed med in last 2 wks? - missed 3 to 5 days | 0 | 0
  Week 4: 01. Missed med in last 2 wks? - missed once/twice | 1 | 4
  Week 4: 01. Missed med in last 2 wks? - No, took every day | 6 | 2
  Week 4: 02a. Stopped med during last 2 wks? - Yes | 0 | 1
  Week 4: 02a. Stopped med during last 2 wks? - No | 7 | 6
  Week 4: 2aii. Stopped meds due to: Side effects - Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 4: 2aii. Stopped meds due to: Symptoms increase -Yes | NA — This follow-up item was not administered for this group and timepoint. | 1
  Week 4: 2aii. Stopped meds due to: Symptoms decrease -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 4: 2aii. Stopped meds due to: Ran out of meds -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 4: 2aii. Stopped meds due to: Forgot to take -Yes | NA — This follow-up item was not administered for this group and timepoint. | 1
  Week 4: 02b. Skipped med in last 2 wks? - Yes | 0 | 4
  Week 4: 02b. Skipped med in last 2 wks? - No | 7 | 3
  Week 4: 02bi. Skipped meds due to: Side effects - Yes | NA — This follow-up item was not administered for this group and timepoint. | 1
  Week 4: 02bi. Skipped meds due to: Symptoms increase -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 4: 02bi. Skipped meds due to: Symptoms decrease -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 4: 02bi. Skipped meds due to: Ran out of meds -Yes | NA — This follow-up item was not administered for this group and timepoint. | 1
  Week 4: 02bi. Skipped meds due to: Forgot to take -Yes | NA — This follow-up item was not administered for this group and timepoint. | 3
  Week 4: 02bi. Skipped meds due to: Other reason -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 4: 02c. Have you reduced med dosage? - Yes | 0 | 0
  Week 4: 02c. Have you reduced med dosage? - No | 7 | 7
  Week 4: 02ci. Reduced meds due to: Side effects - Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 4: 02ci. Reduced meds due to: Symptoms increase -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 4: 02ci. Reduced meds due to: Symptoms decrease -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 4: 02ci. Reduced meds due to: Ran out of meds -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 4: 02ci. Reduced meds due to: Forgot to take -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 4: 02ci. Reduced meds due to: Other reason -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 4: 02d. Have you increased med dosage? - Yes | 1 | 2
  Week 4: 02d. Have you increased med dosage? - No | 6 | 5
  Week 4: 02di. Increased meds due to: Side effects - Yes | 0 | 0
  Week 4: 02di.Increased meds due to: Symptoms increase -Yes | 1 | 0
  Week 4: 02di.Increased meds due to: Symptoms decrease -Yes | 0 | 0
  Week 4: 02di.Increased meds due to: Ran out of meds -Yes | 0 | 0
  Week 4: 02di.Increased meds due to: Forgot to take -Yes | 0 | 0
  Week 4: 02di.Increased meds due to: Other reason -Yes | 0 | 2
  Week 4: 02ai. Stopped meds 3 days ago | NA — This follow-up item was not administered for this group and timepoint. | 1
  Week 4: 02ai. Stopped meds 14 days ago | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 4: 02ai. Stopped meds 2 ± 0 days days ago | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 8: 01. Missed med in last 2 wks? - missed all 14 days | 0 | 1
  Week 8: 01. Missed med in last 2 wks? - missed 6 to 8 days | 0 | 0
  Week 8: 01. Missed med in last 2 wks? - missed 3 to 5 days | 1 | 1
  Week 8: 01. Missed med in last 2 wks? - missed once/twice | 0 | 3
  Week 8: 01. Missed med in last 2 wks? - No, took every day | 4 | 2
  Week 8: 02a. Stopped med during last 2 wks? - Yes | 0 | 1
  Week 8: 02a. Stopped med during last 2 wks? - No | 5 | 6
  Week 8: 2aii. Stopped meds due to: Side effects - Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 8: 2aii. Stopped meds due to: Symptoms increase -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 8: 2aii. Stopped meds due to: Symptoms decrease -Yes | NA — This follow-up item was not administered for this group and timepoint. | 1
  Week 8: 2aii. Stopped meds due to: Ran out of meds -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 8: 2aii. Stopped meds due to: Forgot to take -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 8: 02b. Skipped med in last 2 wks? - Yes | 1 | 3
  Week 8: 02b. Skipped med in last 2 wks? - No | 4 | 4
  Week 8: 02bi. Skipped meds due to: Side effects - Yes | 0 | 0
  Week 8: 02bi. Skipped meds due to: Symptoms increase -Yes | 0 | 0
  Week 8: 02bi. Skipped meds due to: Symptoms decrease -Yes | 0 | 0
  Week 8: 02bi. Skipped meds due to: Ran out of meds -Yes | 0 | 1
  Week 8: 02bi. Skipped meds due to: Forgot to take -Yes | 0 | 2
  Week 8: 02bi. Skipped meds due to: Other reason -Yes | 1 | 0
  Week 8: 02c. Have you reduced med dosage? - Yes | 1 | 1
  Week 8: 02c. Have you reduced med dosage? - No | 4 | 6
  Week 8: 02ci. Reduced meds due to: Side effects - Yes | 0 | 0
  Week 8: 02ci. Reduced meds due to: Symptoms increase -Yes | 0 | 0
  Week 8: 02ci. Reduced meds due to: Symptoms decrease -Yes | 0 | 1
  Week 8: 02ci. Reduced meds due to: Ran out of meds -Yes | 0 | 0
  Week 8: 02ci. Reduced meds due to: Forgot to take -Yes | 0 | 0
  Week 8: 02ci. Reduced meds due to: Other reason -Yes | 1 | 0
  Week 8: 02d. Have you increased med dosage? - Yes | 0 | 0
  Week 8: 02d. Have you increased med dosage? - No | 5 | 7
  Week 8: 02di. Increased meds due to: Side effects - Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 8: 02di.Increased meds due to: Symptoms increase -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 8: 02di.Increased meds due to: Symptoms decrease -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 8: 02di.Increased meds due to: Ran out of meds -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 8: 02di.Increased meds due to: Forgot to take -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 8: 02di.Increased meds due to: Other reason -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 8: 02ai. Stopped meds 3 days ago | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 8: 02ai. Stopped meds 14 days ago | NA — This follow-up item was not administered for this group and timepoint. | 1
  Week 8: 02ai. Stopped meds 2 ± 0 days days ago | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 12: 01. Missed med in last 2 wks? - missed all 14 days | 0 | 1
  Week 12: 01. Missed med in last 2 wks? - missed 6 to 8 days | 1 | 0
  Week 12: 01. Missed med in last 2 wks? - missed 3 to 5 days | 0 | 1
  Week 12: 01. Missed med in last 2 wks? - missed once/twice | 1 | 3
  Week 12: 01. Missed med in last 2 wks? - No, took every day | 3 | 2
  Week 12: 02a. Stopped med during last 2 wks? - Yes | 0 | 2
  Week 12: 02a. Stopped med during last 2 wks? - No | 5 | 5
  Week 12: 2aii. Stopped meds due to: Side effects - Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 12: 2aii. Stopped meds due to: Symptoms increase -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 12: 2aii. Stopped meds due to: Symptoms decrease -Yes | NA — This follow-up item was not administered for this group and timepoint. | 1
  Week 12: 2aii. Stopped meds due to: Ran out of meds -Yes | NA — This follow-up item was not administered for this group and timepoint. | 1
  Week 12: 2aii. Stopped meds due to: Forgot to take -Yes | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 12: 02b. Skipped med in last 2 wks? - Yes | 1 | 2
  Week 12: 02b. Skipped med in last 2 wks? - No | 4 | 5
  Week 12: 02bi. Skipped meds due to: Side effects - Yes | 0 | 0
  Week 12: 02bi. Skipped meds due to: Symptoms increase -Yes | 0 | 0
  Week 12: 02bi. Skipped meds due to: Symptoms decrease -Yes | 0 | 0
  Week 12: 02bi. Skipped meds due to: Ran out of meds -Yes | 0 | 1
  Week 12: 02bi. Skipped meds due to: Forgot to take -Yes | 1 | 1
  Week 12: 02bi. Skipped meds due to: Other reason -Yes | 0 | 0
  Week 12: 02c. Have you reduced med dosage? - Yes | 1 | 0
  Week 12: 02c. Have you reduced med dosage? - No | 4 | 7
  Week 12: 02ci. Reduced meds due to: Side effects - Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02ci. Reduced meds due to: Symptoms increase -Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02ci. Reduced meds due to: Symptoms decrease -Yes | 1 | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02ci. Reduced meds due to: Ran out of meds -Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02ci. Reduced meds due to: Forgot to take -Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02ci. Reduced meds due to: Other reason -Yes | 0 | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02d. Have you increased med dosage? - Yes | 0 | 0
  Week 12: 02d. Have you increased med dosage? - No | 5 | 7
  Week 12: 02di. Increased meds due to: Side effects - Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02di.Increased meds due to: Symptoms increase -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02di.Increased meds due to: Symptoms decrease -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02di.Increased meds due to: Ran out of meds -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02di.Increased meds due to: Forgot to take -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02di.Increased meds due to: Other reason -Yes | NA — This follow-up item was not administered for this group and timepoint. | NA — This follow-up item was not administered for this group and timepoint.
  Week 12: 02ai. Stopped meds 3 days ago | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 12: 02ai. Stopped meds 14 days ago | NA — This follow-up item was not administered for this group and timepoint. | 0
  Week 12: 02ai. Stopped meds 2 ± 0 days days ago | NA — This follow-up item was not administered for this group and timepoint. | 2

2. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 measures degree of depression severity. Possible range of scores for the PHQ-9 is 0-27. Higher values represent a worse outcome. Specifically, scores of 0-4 indicate minimal or no depression; 5-9 is mild; 10-14 is moderate; 15-19 is moderately severe; and 20-27 is severe.
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MedLink System | Treatment As Usual
Number analyzed (Participants) | 8 | 7
units on a scale
  Baseline | 15.25 (6.07) | 11.43 (2.15)
  Week 4 | 10.57 (8.64) | 5.57 (2.94)
  Week 8 | 5.80 (4.55) | 3.43 (2.51)
  Week 12 | 5.20 (2.39) | 2.00 (2.24)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | MedLink System | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes